CLINICAL TRIAL: NCT03319862
Title: Post-massive Weight Loss Chest Contouring: Inferior Pedicle Technique in Pseudo-gynecomastia Correction
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PEDINF
Record Dates: First submitted 2017-10-16; First posted 2017-10-24 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2017-10

CONDITIONS: Gynecomastia
MeSH Terms: conditions — Gynecomastia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Inferior pédicule gynaecomastia — Inferior pédicule gynaecomastia

SUMMARY:
The massive weight loss leads an important excess of skin on thoracic level giving the aspect of a feminine breast with a relatively important ptose. Several techniques were described in the literature about gynaecomastia , but the post-bariatric pseudo-gynaecomastia was not handled yet enough. Moreover, there is no single consensual technique on this subject. The technique used in this service was described for the first time in 2008 ( 1 ) on a serie of 8 patients with an average follow-up of 13 months. Although the results are promising, no other publication was done, and the procedure remains badly represented in the world literature.

ELIGIBILITY:
Inclusion Criteria:

* inferior pedicle gynaecomastia surgery
* Age > 16

Exclusion Criteria:

* Age < 16

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: every patient hospitalized for gynaecomastia but only whose have a inferior pedicle gynaecomastia are selected for the project.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
aesthetic result score | Average of 6 months post-surgery
  patient answer to a satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philippe LEVAN, MD, Study Director — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France